CLINICAL TRIAL: NCT02547714
Title: A Multi-center, Open-label Study of Subcutaneous Secukinumab to Evaluate Efficacy and Safety for 16 Weeks in Patients With Plaque Psoriasis Who Had Inadequate Response to Cyclosporine A
Brief Title: Open-label Study of Subcutaneous Secukinumab to Evaluate Efficacy and Safety in Patients With Plaque Psoriasis Who Had Inadequate Response to Cyclosporine A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457AJP01
Record Dates: First submitted 2015-07-12; First posted 2015-09-11 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-08

CONDITIONS: Plaque Psoriasis
Keywords: cyclosporine A
MeSH Terms: interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Secukinumab (AIN457) 300 mg (Experimental): Participants received secukinumab 300 mg subcutaneously (s.c.) (two 150 mg injections) on Day 1 and at Weeks 1, 2, 3, 4, 8 and 12.
  Interventions: Drug: Secukinumab (AIN457)

INTERVENTIONS:
Drug: Secukinumab (AIN457) — Secukinumab was supplied as 150 mg doses, provided in 1 mL prefilled syringes.

SUMMARY:
The purpose of this study was to assess the efficacy and safety of secukinumab at Week 16 based on psoriasis area and severity index (PASI) 75 in subjects who had inadequate response to cyclosporine A.

ELIGIBILITY:
Inclusion criteria:

* Plaque psoriasis diagnosed for at least 6 months before baseline - Treated with cyclosporine A for at least 12 weeks prior to baseline
* Currently treated with cyclosporine A at baseline for psoriasis but is a primary or secondary inadequate response as defined at baseline by:

  * PASI score of 10 or greater and
  * IGA mod 2011 score of 2 or greater (based on a scale of 0 to 4)

Exclusion Criteria:

* Forms of psoriasis other than plaque (e.g., pustular, erythrodermic and guttate psoriasis). -Drug-induced psoriasis (i.e., new onset or current exacerbation from beta-blockers, calcium channel blockers or lithium).
* Patients who have to discontinue cyclosporine A treatment due to side effects like renal impairment (serum creatinine exceeding 176.8 μmol/L [2.0 mg/dL]) and hypertension at screening.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-06-16 (Actual); Primary Completion 2016-05-02 (Actual); Study Completion 2016-05-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- Japan (10):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-Ku, Tokyo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The overall treatment period consisted of a 4 week induction period (Day 1 and weeks 1, 2, 3 and 4) and a 12 week maintenance period (weeks 8 and 12). All participants entered and completed both periods.
Period: Overall Study
Arm/Group | Secukinumab (AIN457) 300 mg
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Secukinumab (AIN457) 300 mg
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.5 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved ≥ 75% Psoriasis Area and Severity Index (PASI 75)
Description: PASI is a combined assessment of a lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). The body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for a final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area * area score weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4). PASI 75 was defined as participants achieving >= 75% improvement from baseline.
Time Frame: Week 16
Population: The full analysis set, which included all participants who received at least one dose of study drug, was analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab (AIN457) 300 mg
Number analyzed (Participants) | 34
Percentage of participants | 82.4

2. Secondary Outcome: Mean Percent Change From Baseline in PASI Score
Description: PASI is a combined assessment of a lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). The body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for a final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area * area score weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4). A negative change from baseline indicates improvement.
Time Frame: Week 4
Population: The full analysis set, which included all participants who received at least one dose of study drug, was analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Secukinumab (AIN457) 300 mg
Number analyzed (Participants) | 34
Percent change | -65.64 (37.200)

3. Secondary Outcome: Percentage of Participants Achieving PASI 50 or PASI 75
Description: PASI is a combined assessment of a lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). The body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for a final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area * area score weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4).
  PASI 50 and PASI 75 were defined as participants achieving >= 50% or >= 75% improvement from baseline, respectively.
Time Frame: Week 4
Population: The full analysis set, which included all participants who received at least one dose of study drug, was analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab (AIN457) 300 mg
Number analyzed (Participants) | 34
Percentage of participants
  PASI 50 | 76.5
  PASI 75 | 44.1

4. Secondary Outcome: Percentage of Participants Achieving PASI 90 and Investigator's Global Assessment (IGA) of 0 or 1 Response
Description: PASI is a combined assessment of a lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). The body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for a final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area * area score weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4).
  PASI 90 was defined as participants achieving >= 90% improvement from baseline. The IGA scale is static, i.e. it referred exclusively to the participant's disease at the time of assessment and did not compare with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe.
Time Frame: Week 16
Population: The full analysis set, which included all participants who received at least one dose of study drug, was analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab (AIN457) 300 mg
Number analyzed (Participants) | 34
Percentage of participants
  PASI 90 | 64.7
  IGA 0/1 | 70.6

5. Secondary Outcome: Mean Percent Change From Baseline in Dermatology Life Quality Index (DLQI) Score
Description: The DLQI is a ten item general dermatology disability index designed to assess health-related quality of life in adult participants with skin diseases such as eczema, psoriasis, acne and viral warts. It is a self-administered questionnaire which includes domains of daily activity, leisure, personal relationships, symptoms and feelings, treatment and school/work activities. Each domain has 4 response categories ranging from 0 (not at all) to 3 (very much). "Not relevant" is a valid score also and is scored as 0. The DLQI total score is a sum of all 10 responses. Scores range from 0 to 30 with higher scores indicating greater health-related quality of life impairment. A negative mean percentage change from baseline indicates improvement.
Time Frame: Week 16
Population: The full analysis set was considered for the analysis. Only participants who had both baseline and week 16 values were included in the analysis. The full analysis set included all participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Secukinumab (AIN457) 300 mg
Number analyzed (Participants) | 33
Percent change | -63.07 (59.192)

6. Secondary Outcome: Percentage of Participants Achieving DLQI 0 or 1
Description: The DLQI is a ten item general dermatology disability index designed to assess health-related quality of life in adult participants with skin diseases such as eczema, psoriasis, acne and viral warts. It is a self-administered questionnaire which includes domains of daily activity, leisure, personal relationships, symptoms and feelings, treatment and school/work activities. Each domain has 4 response categories ranging from 0 (not at all) to 3 (very much). "Not relevant" is a valid score also and is scored as 0. The DLQI total score is a sum of all 10 responses. Scores range from 0 to 30 with higher scores indicating greater health-related quality of life impairment.
Time Frame: Week 16
Population: The full analysis set, which included all participants who received at least one dose of study drug, was analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Secukinumab (AIN457) 300 mg
Number analyzed (Participants) | 34
Percentage of participants | 76.5

ADVERSE EVENTS:
Groups:
- Entire Period - Secukinumab (AIN457): Participants received secukinumab 300 mg subcutaneously (s.c.) (two 150 mg injections) on Day 1 and at Weeks 1, 2, 3, 4, 8 and 12.
- Induction Period - Secukinumab (AIN457): During the induction period, participants received secukinumab 300 mg subcutaneously (s.c.) (two 150 mg injections) on Day 1 and at Weeks 1, 2, 3, and 4.
Arm/Group | Entire Period - Secukinumab (AIN457) | Induction Period - Secukinumab (AIN457)
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 24/34 | 10/34
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Entire Period - Secukinumab (AIN457) (N=34) | Induction Period - Secukinumab (AIN457) (N=34)
Conjunctivitis allergic (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Injection site erythema (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Angular cheilitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 7 | 4
Paronychia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1
Tinea versicolour (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Hot flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.